CLINICAL TRIAL: NCT02739893
Title: Randomized Trial Comparing the Usefulness of A Scope Guide Assisted Colonoscopy Versus Conventional Colonoscopy
Brief Title: Usefulness of A Scope Guide Assisted Colonoscopy Versus Conventional Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Shajan P. Sugandha, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: F141223002
Record Dates: First submitted 2016-03-25; First posted 2016-04-15 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Colonoscopy, Colorectal
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scope Guide Assisted (Experimental): Scope Guide Assist to be utilized during colonoscopy
  Interventions: Procedure: Scope Guide Assist
- Standard (Placebo Comparator): Colonoscopy completed using current SOC without scopeguide assist.
  Interventions: Procedure: Standard procedure for colonoscopy

INTERVENTIONS:
Procedure: Scope Guide Assist — Olympus has developed a new instrument which provides physicians a real-time, three dimensional visualization of position and configuration during colonoscopy. The Olympus ScopeGuide technology has received FDA clearance and can be used within the United States. The new technology called the 'scopeguide' has been developed that uses magnetic coils embedded into the scope to create a 3 D image of the shape of the entire scope inside the body that is projected onto the monitor to see. This acts as a "GPS" and shows the advancement of the scope through bends providing information on loops and thereby eliminating chances of loop formation, helping in loop reduction and also reducing the number of external maneuvers that may be required for the completion of colonoscopy.
  Arms: Scope Guide Assisted
Procedure: Standard procedure for colonoscopy
  Arms: Standard

SUMMARY:
The aim of this study is to see if use of ScopeGuide, as compared to the traditional colonoscope, improves successful completion of colonoscopy procedures as evaluated by ease of completion, time to completion, and reduction in the number of mechanical loops and external maneuvers required to advance the scope. Other outcome measures include looking at the amount of sedation required (independent of weight) and polyp rate detection.

DETAILED DESCRIPTION:
Currently, the standard practice consists of utilizing a traditional colonoscope and depends on manual manipulation and learned expertise of human anatomy. If the scope guide reduces the amount of external maneuvers required, this will reduce patient discomfort and may reduce sedative requirements during procedure. Reduction in mechanical loops formed while advancing the scope will reduce the amount of time per procedure and potentially increase polyp detection. Additionally, if the physician is unable to complete the procedure (as indicated by reaching the cecum (anatomical structure signifying the end of the colon), clinical data may be lost. A reduction in the number of loops formed and ease of advancing scope will facilitate completion of procedure.

The patient will not be exposed to any inconvenience, danger, or discomfort as a result of study participation. Patients undergoing colonoscopy as SOC, if enrolled into the study, will be randomized by envelope at the time of procedure. If the patient is randomized to the scope guide, the PI simply activates the guide through a mechanical button placed on the scope itself. If the patient is randomized to SOC, the physician proceeds with the colonoscopy without activating the scope guide. The same scope is used regardless of randomization result. The physician is able to turn on and off the magnetic function through the touch of a button.

The colonoscopy procedure itself is not dependent upon use of the scope guide. However, the use of the scope guide may assist the physician in performing the procedure with less physical manipulation. Without the use of the ScopeGuide, an endoscopist is able to perform the procedure based off anatomical knowledge and through the use of maneuvers such as changing the patient position and applying external pressure. This study will test if the ScopeGuide decreases the number of maneuvers required for completion. If the number of maneuvers is decreased, it is likely to decrease patient discomfort and decrease the duration of procedure. This study will also test of the ScopeGuide increases completeness of procedure.

300 patients undergoing SOC colonoscopy will be randomized 1:1 to receive traditional colonoscopy or scope guide assisted colonoscopy.

This study will assess if the scope guide assist function improves successful completion of colonoscopy, time to completion, and reduction in the number of mechanical loops and external maneuvers required to advance the scope. Polyp detection rate and amount of sedation required will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* able to safely undergo colonoscopy without history of colorectal surgery, colonic stricture or obstruction.

Exclusion Criteria:

* history of colorectal surgery,
* current colonic stricture or obstruction,
* unable to safely undergo colonoscopy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Mean cecum intubation time for each arm | from start of colonoscopy until completion - approximately 60 minutes
  time in minutes to reach cecum destination in each arm
Mean time in minutes to complete colonoscopy | from start of colonoscopy until completion - approximately 60 minutes
  Mean time to completion for each arm
Mean number of mechanical loops required to complete procedure for each arm | from start of colonoscopy until completion - approximately 60 minutes
  Each mechanical loop will be counted as 1 (one)
Number of mean external maneuvers per procedure between groups | from start of colonoscopy until completion - approximately 60 minutes
  mean number of external maneuvers across all subjects in each arm

SECONDARY OUTCOMES:
Mean amount of sedation per arm | from start of colonoscopy until completion - approximately 60 minutes
  amount of sedation in mg per arm
Percent of subjects with detectable polyps per arm | from start of colonoscopy until completion - approximately 60 minutes
  percent of subjects in each with at least identifiable polyp

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Birmingham, Alabama, United States